CLINICAL TRIAL: NCT01751724
Title: Use of Caffeine to Reduce Length of Mechanical Ventilation in Preterm Infants
Brief Title: Caffeine to Reduce Mechanical Ventilation in Preterm Infants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Safety
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Eduardo Bancalari, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20120786
Record Dates: First submitted 2012-12-12; First posted 2012-12-18 (Estimated); Results first posted 2017-06-19 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-05

CONDITIONS: Prematurity; Apnea; Respiratory Failure
Keywords: Premature infants; Caffeine; Methylxanthines; Mechanical ventilation; Oxygen; Weaning; Bronchopulmonary dysplasia
MeSH Terms: conditions — Premature Birth; Apnea; Respiratory Insufficiency; Bronchopulmonary Dysplasia | interventions — caffeine citrate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Caffeine Arm (Experimental): Subjects randomized to this arm will receive blinded Caffeine citrate.
  Interventions: Drug: Caffeine citrate
- Placebo Arm (Placebo Comparator): Subjects randomized to this arm will receive blinded Placebo (equivalent volume of normal saline).
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: Caffeine citrate — Enrolled subjects will be randomized to receive a study drug consisting of either blinded Caffeine citrate.
  Randomization and study drug preparation will be done by the NICU pharmacy. Investigators and clinicians will be blinded to the assigned drug.
  After randomization, an initial loading dose of 20 mg/Kg of study drug will be followed by a 5 mg/Kg/day maintenance dose. The assigned study drug will be administered intravenous or orally as determined by the clinical team.
  Infants will continue to receive the study drug until 12 hours prior to the first elective extubation.
  Arms: Caffeine Arm
Other: Normal saline — Enrolled subjects will be randomized to receive a study drug consisting of blinded Placebo (equivalent volume of normal saline).
  Randomization and study drug preparation will be done by the NICU pharmacy. Investigators and clinicians will be blinded to the assigned drug.
  After randomization, an initial loading dose of 20 mg/Kg of study drug will be followed by a 5 mg/Kg/day maintenance dose. The assigned study drug will be administered intravenous or orally as determined by the clinical team.
  Infants will continue to receive the study drug until 12 hours prior to the first elective extubation.
  Arms: Placebo Arm

SUMMARY:
Most premature infants require mechanical ventilation for prolonged periods of time and a significant proportion of them develop Bronchopulmonary Dysplasia (BPD). Caffeine is a stimulant of the respiratory center and has been used for the treatment of Apnea of Prematurity in infants not requiring mechanical ventilation or to facilitate weaning from mechanical ventilation by starting therapy shortly before extubation. Recently the use of Caffeine in ventilated infants has been initiated earlier because of the reported reduction in BPD. However there is paucity of data supporting this practice.

Because protracted mechanical ventilation and supplemental oxygen increase the risk of developing BPD, a therapy that would facilitate the reduction of the respiratory support and shorten its duration is desirable. Therefore, it is of importance to evaluate the effects of early Caffeine initiation and administration during the course of mechanical ventilation in preterm infants by means of a randomized placebo-controlled trial.

Hypothesis:

The primary hypothesis of this study is that early use of caffeine in mechanically ventilated preterm infants will reduce the time to first elective extubation and secondarily, that this will reduce the total duration of mechanical ventilation and oxygen supplementation, and reduce the incidence and severity of BPD.

Objective:

The objective of this trial is to evaluate the effects of early caffeine use during mechanical ventilation on the time to first elective extubation, total duration of mechanical ventilation and oxygen supplementation, and the incidence of BPD.

Study Design:

This will be a single-center prospective, randomized, double-blind, placebo controlled clinical trial.

Population:

Premature neonates born between 23 and 30 completed weeks of gestation, who require mechanical ventilation within the first 5 days of life will be enrolled. Infants with major congenital anomalies or small for gestational age will be excluded.

Methods:

Infants will be randomized within the first 5 days to receive a study drug consisting of either blinded Caffeine citrate or blinded Placebo (equivalent volume of normal saline). Infants will continue to receive the study drug until the first elective extubation.

ELIGIBILITY:
Inclusion Criteria:

* Premature neonates born between 23 and 30 completed weeks of gestation.
* Requiring mechanical ventilation within the first 5 postnatal days
* Written-informed parental consent for the study

Exclusion Criteria:

* Major congenital anomalies
* Small for gestational age

Ages: 1 Day to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2012-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Bancalari, M.D., Principal Investigator — University of Miami; Nelson Claure, M.Sc., Ph.D., Principal Investigator — University of Miami
Locations (1):
- NICU, Holtz Children's Hospital, Jackson Health System, Miami, Florida, United States

REFERENCES:
- [Derived] Amaro CM, Bello JA, Jain D, Ramnath A, D'Ugard C, Vanbuskirk S, Bancalari E, Claure N. Early Caffeine and Weaning from Mechanical Ventilation in Preterm Infants: A Randomized, Placebo-Controlled Trial. J Pediatr. 2018 May;196:52-57. doi: 10.1016/j.jpeds.2018.01.010. Epub 2018 Mar 6. PMID 29519541

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted at the Holtz Children's Hospital newborn intensive care unit of Jackson Health System/University of Miami Medical Center from January 2013 to October 2015.
Pre-assignment Details: 87 infants were enrolled. Of these, 1 died before randomization. 86 infants were randomized and assigned an intervention arm.
Groups:
- Caffeine Arm: Subjects randomized to this arm will receive blinded Caffeine citrate.
  Caffeine citrate: Enrolled subjects will be randomized to receive a study drug consisting of either blinded Caffeine citrate.
  Randomization and study drug preparation will be done by the NICU pharmacy. Investigators and clinicians will be blinded to the assigned drug.
  After randomization, an initial loading dose of 20 mg/Kg of study drug will be followed by a 5 mg/Kg/day maintenance dose. The assigned study drug will be administered intravenous or orally as determined by the clinical team.
  Infants will continue to receive the study drug until 12 hours prior to the first elective extubation.
- Placebo Arm: Subjects randomized to this arm will receive blinded Placebo (equivalent volume of normal saline).
  Normal saline: Enrolled subjects will be randomized to receive a study drug consisting of blinded Placebo (equivalent volume of normal saline).
  Randomization and study drug preparation will be done by the NICU pharmacy. Investigators and clinicians will be blinded to the assigned drug.
  After randomization, an initial loading dose of 20 mg/Kg of study drug will be followed by a 5 mg/Kg/day maintenance dose. The assigned study drug will be administered intravenous or orally as determined by the clinical team.
  Infants will continue to receive the study drug until 12 hours prior to the first elective extubation.
Period: Overall Study
Arm/Group | Caffeine Arm | Placebo Arm
Started | 42 | 44
Completed | 41 | 42
Not Completed | 1 | 2
Not completed — extubated bef.start assigned treatment | 1 | 0
Not completed — withdrawn by parent | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caffeine Arm | Placebo Arm | Total
Number analyzed (Participants) | 41 | 42 | 83
Age, Continuous [Mean (Standard Deviation); unit: hours] | 48 (25) | 49 (31) | 48 (28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 25 | 36
  Male | 30 | 17 | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black race | 19 | 21 | 40
Gestational age [Median (Inter-Quartile Range); unit: weeks] | 25.7 [24.3 to 27.0] | 26.1 [24.2 to 28.4] | 25.9 [24.2 to 27.5]
Birth weight [Median (Inter-Quartile Range); unit: grams] | 670 [605 to 915] | 720 [643 to 894] | 700 [615 to 906]
Fraction of inspired oxygen at enrollment [Median (Inter-Quartile Range); unit: oxygen fraction] | 0.25 [0.21 to 0.37] | 0.23 [.21 to .30] | .24 [.21 to .33]
Mean airway pressure at enrollment [Median (Inter-Quartile Range); unit: centimeters of water] | 9 [8 to 11] | 8 [8 to 10] | 9 [8 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Age at First Successful Extubation
Description: Defined as age of extubation with infant remaining extubated for more than 24 hours.
Time Frame: From birth to until 36 weeks postmenstrual age
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Caffeine Arm | Placebo Arm
Number analyzed (Participants) | 41 | 42
days | 24 [9.5 to 41] | 20 [9.3 to 43]

2. Secondary Outcome: Survival
Time Frame: From the time of randomization up to 36 weeks corrected age, or until the time of discharge or death
Measure: Count of Participants; unit: Participants
Arm/Group | Caffeine Arm | Placebo Arm
Number analyzed (Participants) | 41 | 42
Participants | 32 | 37

3. Secondary Outcome: Total Duration of Mechanical Ventilation
Time Frame: From the time of first intubation until the last extubation, up to 36 weeks corrected age
Population: Infants alive at 36 weeks postmenstrual age
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Caffeine Arm | Placebo Arm
Number analyzed (Participants) | 32 | 37
days | 32 [11 to 43] | 26 [10 to 44]

4. Secondary Outcome: Total Duration of Oxygen Supplementation
Time Frame: From the time of first initiation until the last day of oxygen supplementation, up to 36 weeks corrected age
Population: Infants alive at 36 weeks postmenstrual age
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Caffeine Arm | Placebo Arm
Number analyzed (Participants) | 32 | 37
days | 55 [31 to 86] | 59 [36 to 106]

5. Secondary Outcome: Number of Infants With Bronchopulmonary Dysplasia (BPD)
Description: BPD defined as need for oxygen for at least 28 days and at 36 weeks post-menstrual age.
Time Frame: Evaluated at 36 weeks corrected postmenstrual age
Population: Infants alive at 36 weeks postmenstrual age
Measure: Count of Participants; unit: Participants
Arm/Group | Caffeine Arm | Placebo Arm
Number analyzed (Participants) | 32 | 37
Participants | 15 | 20

6. Secondary Outcome: Survival Without BPD
Description: Discharge alive without BPD. BPD defined as need for oxygen for at least 28 days and at 36 weeks post-menstrual age.
Time Frame: From the time of randomization until 36 weeks corrected age, discharge or death
Measure: Count of Participants; unit: Participants
Arm/Group | Caffeine Arm | Placebo Arm
Number analyzed (Participants) | 41 | 42
Participants | 18 | 18

7. Other Pre Specified Outcome: Number of Infants With Pulmonary Hemorrhage
Time Frame: From enrollment until 36 weeks postmenstrual age, discharge or death
Measure: Count of Participants; unit: Participants
Arm/Group | Caffeine Arm | Placebo Arm
Number analyzed (Participants) | 41 | 42
Participants | 7 | 4

8. Other Pre Specified Outcome: Number of Infants With Necrotizing Enterocolitis
Time Frame: From enrollment until 36 weeks postmenstrual age, discharge or death
Measure: Count of Participants; unit: Participants
Arm/Group | Caffeine Arm | Placebo Arm
Number analyzed (Participants) | 41 | 42
Participants | 7 | 2

9. Other Pre Specified Outcome: Number of Infants With Septicemia
Description: Septicemia defined as positive blood culture
Time Frame: From enrollment until 36 weeks postmenstrual age, discharge or death
Measure: Count of Participants; unit: Participants
Arm/Group | Caffeine Arm | Placebo Arm
Number analyzed (Participants) | 41 | 42
Participants | 12 | 10

10. Other Pre Specified Outcome: Number of Infants With Severe Intraventricular Hemorrhage
Description: Severe intraventricular hemorrhage defined as grade III or higher
Time Frame: From enrollment until 36 weeks postmenstrual age, discharge or death
Measure: Count of Participants; unit: Participants
Arm/Group | Caffeine Arm | Placebo Arm
Number analyzed (Participants) | 41 | 42
Participants | 12 | 6

11. Other Pre Specified Outcome: Number of Infants With Severe Retinopathy of Prematurity
Description: Severe retinopathy of prematurity defined as stage 3 or higher
Time Frame: From enrollment until 36 weeks postmenstrual age, discharge or death
Measure: Count of Participants; unit: Participants
Arm/Group | Caffeine Arm | Placebo Arm
Number analyzed (Participants) | 41 | 42
Participants | 3 | 5

ADVERSE EVENTS:
Arm/Group | Caffeine Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 9/41 | 5/42
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/42
Other Adverse Events (participants affected / at risk) | 0/41 | 0/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caffeine Arm (N=41) | Placebo Arm (N=42)
Seizures (Nervous system disorders) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No